CLINICAL TRIAL: NCT03873038
Title: Single and Multiple Dose Clinical Trial to Study the Safety and Pharmacokinetics of MK-2060 in Older Participants With End-Stage Renal Disease on Hemodialysis
Brief Title: Safety and Pharmacokinetics of MK-2060 in Older Participants With End-Stage Renal Disease on Hemodialysis (MK-2060-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 2060-004; MK-2060-004 (Other: Merck)
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Renal Dialysis; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Panel A- MK-2060 (8 mg) (Experimental): Participants will receive a single 8-mg dose of MK-2060 via intravenous (IV) infusion.
  Interventions: Drug: MK-2060
- Part 1: Panel B- MK-2060 (20 mg) (Experimental): Participants will receive a single 20-mg dose of MK-2060 via IV infusion.
  Interventions: Drug: MK-2060
- Part 1: Panel C- MK-2060 (40 mg) (Experimental): Participants will receive a single 40-mg dose of MK-2060 via IV infusion.
  Interventions: Drug: MK-2060
- Part 1: Placebo (Placebo Comparator): Participants will receive a single dose of placebo via IV infusion.
  Interventions: Drug: Placebo
- Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance (Experimental): Participants will receive three doses of up to 25 mg MK-2060 via IV infusion in the first week (Week 1), followed by a single dose of up to 25 mg MK-2060 via IV infusion weekly for 3 weeks (Weeks 2-4)
  Interventions: Drug: MK-2060
- Part 2: Placebo (Placebo Comparator): Participants will receive three doses of placebo via IV infusion in the first week and then a single dose of placebo via IV infusion weekly for 3 weeks (Weeks 2-4)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-2060 — Part 1: Single doses (8 mg, 20 mg, or 40 mg) of MK-2060 will be administered via IV infusion on Day 1.
  Part 2: Three doses of 25 mg of MK- 2060 administered via IV infusion on Days 1, 3 and 5; Followed by single doses of 25 mg of MK-2060 administered via IV infusion on Days 8, 15, and 22.
  Arms: Part 1: Panel A- MK-2060 (8 mg); Part 1: Panel B- MK-2060 (20 mg); Part 1: Panel C- MK-2060 (40 mg); Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance
Drug: Placebo — Part 1: Single dose of placebo will be administered via IV infusion on Day 1. Part 2: Three doses of placebo administered via IV infusion on Days 1, 3 and 5; Followed by single doses of placebo administered via IV infusion on Days 8, 15, and 22.
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of MK-2060 after intravenous (IV) administration of single and multiple doses in older adult participants with end-stage renal disease (ESRD) on hemodialysis (HD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of non-child bearing potential (WONCBP) age ≥40 and ≤80 years for Part 1 and ≥18 and ≤80 years for Part 2.
* End-stage renal disease (ESRD) maintained on stable outpatient hemodialysis (HD) regimen, using an established (> 3 months) and normally functioning, regular flow, uninfected mature arteriovenous (AV) fistula or AV graft and skin consistent with standard chronic HD access injuries, and HD stability defined as ([K, dialyzer clearance, multiplied by t, time, divided by V, patient's total body water] Kt/V) ≥ 1.2 within 3 months prior to dosing at a healthcare center for > 3 months from dosing.
* On HD regimen at least 3 times per week for a minimum of 3 hours per dialysis session, using a complication-free well-maintained AV fistula or AV graft, expected and plan to continue this throughout and for at least 3 months beyond the study.
* Has a Body Mass Index (BMI) ≥ 18 and ≤ 45 kg/m^2, BMI = weight (kg)/height (m)^2.
* Baseline health is judged to be stable based on medical history, physical examination, vital sign measurements and electrocardiogram (ECG) performed prior to randomization.
* Liver function test (serum alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) must be equal to or below 1.5X upper limit of normal (ULN) and deemed not clinically significant by both the investigator and the Sponsor.
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies by agreeing to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant. Also, men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies in that a female participant is eligible to participate if she is not pregnant or breastfeeding and she is not a WOCBP in that she is a postmenopausal female without menses for at least 1 year OR is a surgically sterile female, post hysterectomy, bilateral salpingectomy, oophorectomy or tubal ligation.

Exclusion Criteria:

* Has a history of any clinically significant concomitant disease or condition (including treatment for such conditions) or diseases whose current condition is considered clinically unstable that, in the opinion of the investigator, could either interfere with the study drug, compromise interpretation of study data, or pose an unacceptable risk. Participants with a remote history of uncomplicated medical events (e.g., uncomplicated kidney stones, as defined as spontaneous passage and no recurrence in the last 5 years, or childhood asthma) may be enrolled in the study at the discretion of the investigator.
* Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years. Participants who have had situational depression may be enrolled in the study at the discretion of the investigator.
* Has a history of cancer (malignancy), including adenocarcinoma, with possible exceptions being participants with adequately treated non-melanomatous skin carcinoma; participants with other malignancies which have been successfully treated ≥10 years prior to the pretrial (screening) visit; or participants who, in the opinion of the trial investigator, are highly unlikely to sustain a recurrence for the duration of the trial.
* Has blood coagulation test (activated partial thromboplastin time [aPTT], prothrombin time [PT]) ≥ 20 % outside of normal range on pretrial (screening), which are considered clinically significant by both the investigator and the sponsor.
* Any other clinically significant abnormalities in laboratory test results at screening that would, in the opinion of the investigator, increase the participant's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
* Has a history of deep vein thrombosis or pulmonary embolism. Has a history of vascular access thrombosis within 1 month prior to enrollment. Has a personal or family history of bleeding disorder.
* Has a history of gastrointestinal (GI) bleeding, duodenal polyps or gastric ulcer in the last 5 years or severe hemorrhoidal bleed in last 3 months.
* Has a history of or current frequent epistaxis within the last 3 months or active gingivitis.
* Has ongoing anticoagulant therapy (warfarin, apixaban, dabigatran, rivaroxaban, edoxaban, betrixaban) or antiplatelet therapy (clopidogrel, prasugrel, ticagrelor, ticlopidine). Intradialytic heparin and aspirin are permitted.
* At the time of screening or pre-dose, has planned significant dental procedures (including planned dental surgery), or other planned surgical procedures within duration of participation in the trial.
* Is positive for hepatitis B surface antigen or human immunodeficiency viruses (HIV).
* Has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pre-study (screening) visits.
* Has a history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e. systemic allergic reaction) to prescription or non-prescription drugs or food.
* Has a tattoo, scar, or other physical finding at the area of the infusion site that would interfere with infusion or a local tolerability assessment.
* Has a history of receiving any human immunoglobulin preparation such as intravenous immunoglobulin (IVIG) or RhoGAM within the last year.
* Has a history of receiving any biological therapy (including human blood products or monoclonal antibodies; excluding erythropoietin and insulin) within the last 3 months or 5 half-lives (whichever is longer), or vaccination within the last 1 month (exceptions include seasonal flu vaccine and pneumococcal vaccine within the last month; coronavirus disease 2019 [COVID-19] vaccine that is licensed and approved for emergency use and with the study intervention given 72 hours following vaccination or 48 hours prior to vaccination).
* The exclusion criteria for ECG is a heart rate < 40 or > 110 beats per minute (bpm); corrected Q-T (QTc) interval > 500 minutes/second; any significant arrhythmia or conduction abnormality, (including but not specific to atrioventricular block [2nd degree or higher], Wolff Parkinson White syndrome [unless curative radio ablation therapy]), which, in the opinion of the investigator and sponsor, could interfere with the safety for the individual participant; and non-sustained or sustained ventricular tachycardia (> 2 consecutive ventricular ectopic beats at a rate of > 1.7/second).
* Is unable to refrain from or anticipates the use of medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks prior to administration of the initial dose of study drug, throughout the study until the poststudy visit. Specific allowed and prohibited medications are provided in the protocol.
* Has participated in another investigational study within 4 weeks prior to sponsor's investigational drug (MK-2060/placebo) administration.
* Has a blood pressure >190 mmHg systolic or >110 mmHg diastolic.
* Consumes greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer 354 mL/12 ounces, wine 118 mL/4 ounces, or distilled spirits 29.5 mL/1 ounce) per day. Participants who consume 4 glasses of alcoholic beverages per day may be enrolled at the discretion of the investigator.
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
* Is a regular user of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 2 years. Participants must have a negative serum or saliva drug screen prior to randomization. Participants with a positive drug screen due to the use of physician prescribed medications (e.g., opioids, benzodiazepines, antidepressants) may be enrolled at the discretion of the investigator. In addition, participants with a positive tetrahydrocannabinol (THC) may be enrolled at the discretion of the investigator if the participants' THC use is under 4 times/month and the participants agree to not use during their study participation. Participants with positive THC on screening may have rechecks performed at the discretion of the investigator to ensure compliance with abstinence from THC use during study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - Orlando Clinical Research Center ( Site 0002), Orlando, Florida
  - Prism Research ( Site 0003), Saint Paul, Minnesota
  - New Orleans Center for Clinical Research ( Site 0001), Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and Female of non-childbearing potential (WONCBP) participants with end-stage renal disease (ESRD) on hemodialysis (HD) between the ages of 18 and 80 years (ages ≥ 40 and ≤ 80 for Part 1 and ≥ 18 and ≤ 80 for Part 2) were enrolled in this study.
Groups:
- Part 1: Panel A- MK-2060 (8 mg): Participants received a single 8-mg dose of MK-2060 via intravenous (IV) infusion
- Part 1: Panel B- MK-2060 (20 mg): Participants received a single 20-mg dose of MK-2060 via IV infusion
- Part 1: Panel C- MK-2060 (40 mg): Participants received a single 40-mg dose of MK-2060 via IV infusion
- Part 1: Placebo: Participants received a single dose of placebo via IV infusion
- Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance: Participants received three doses of up to 25 mg MK-2060 via IV infusion in the first week (Week 1), followed by a single dose of up to 25 mg MK-2060 via IV infusion weekly for 3 weeks (Weeks 2-4)
- Part 2: Placebo: Participants received three doses of placebo via IV infusion in the first week and then a single dose of placebo via IV infusion weekly for 3 weeks (Weeks 2-4)
Period: Part 1
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel C- MK-2060 (40 mg) | Part 1: Placebo | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo
Started | 6 | 7 | 6 | 5 | 0 | 0
Completed | 6 | 7 | 6 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel C- MK-2060 (40 mg) | Part 1: Placebo | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo
Started | 0 | 0 | 0 | 0 | 16 (6 participants who received MK-2060 in Part 1 also received MK-2060 in Part 2.) | 5 (One participant who received placebo in Part 1 also received placebo in Part 2.)
Completed | 0 | 0 | 0 | 0 | 15 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Unknon | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Seven participants in Part 1 also participated in Part 2. They have been removed from Part 2 listing and counted only once
Groups:
- Part 1: Panel A- MK-2060 (8 mg): Participants received a single 8-mg dose of MK-2060 via IV infusion
- Total: Total of all reporting groups
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel C- MK-2060 (40 mg) | Part 1: Placebo | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo | Total
Number analyzed (Participants) | 6 | 7 | 6 | 5 | 10 | 4 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (5.1) | 61.1 (4.3) | 58.2 (5.9) | 60.0 (7.3) | 54.7 (7.0) | 52.5 (11.6) | 57.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 2 | 1 | 2 | 0 | 10
  Male | 5 | 3 | 4 | 4 | 8 | 4 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 6 | 5 | 8 | 4 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 3 | 3 | 8 | 4 | 27
  White | 0 | 4 | 3 | 2 | 2 | 0 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Any Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants that experienced an AE was summarized.
Time Frame: Up to 164 days
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Groups:
- Part 1: Panel A- MK-2060 (40 mg): Participants received a single 40-mg dose of MK-2060 via IV infusion
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg) | Part 1: Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 5
Percentage of Participants | 16.7 | 57.1 | 66.7 | 60.0

2. Primary Outcome: Part 2: Percentage of Participants With Any AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experienced an AE was summarized.
Time Frame: Up to 118 days
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo
Number analyzed (Participants) | 16 | 5
Percentage of Participants | 12.5 | 100.0

3. Primary Outcome: Part 1: Percentage of Participants With Any Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants who experienced an SAE was summarized.
Time Frame: Up to 164 days
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg) | Part 1: Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 5
Percentage of Participants | 0.0 | 0.0 | 16.7 | 0.0

4. Primary Outcome: Part 2: Percentage of Participants With Any SAE
Description: An SAE is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants who experienced an SAE was summarized.
Time Frame: Up to 118 days
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo
Number analyzed (Participants) | 16 | 5
Percentage of Participants | 6.3 | 60.0

5. Primary Outcome: Part 1: Percentage of Participants With a Systemic AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The solicited systemic AEs assessed included but not limited to fever, vital sign (VS) changes (tachycardia/hypotension), pruritis, urticarial (hives), lip swelling, angioedema, bronchospasm, stridor, hoarseness, and shortness of breath.
Time Frame: Up to 164 days
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg) | Part 1: Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 5
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: Part 2: Percentage of Participants With a Systemic AE
Description: as for outcome 5
Time Frame: Up to 118 days
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo
Number analyzed (Participants) | 16 | 5
Percentage of Participants | 0.0 | 0.0

7. Primary Outcome: Part 1: Percentage of Participants With an Injection-Site AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The solicited injection-site AEs assessed were pain, tenderness, erythema/redness, and induration/swelling.
Time Frame: Up to 164 days
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg) | Part 1: Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 5
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0

8. Primary Outcome: Part 2: Percentage of Participants With an Injection-Site AE
Description: as for outcome 7
Time Frame: Up to 118 days
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo
Number analyzed (Participants) | 16 | 5
Percentage of Participants | 0.0 | 0.0

9. Primary Outcome: Part 1: Percentage of Participants Discontinuing the Study Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants that discontinued the study due to an AE was summarized.
Time Frame: Up to 164 days
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Groups:
- Part 1: Panel B- MK-2060 (20 mg): Participants received a single 20-mg dose of MK-2060 via IV
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg) | Part 1: Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 5
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0

10. Primary Outcome: Part 2: Percentage of Participants Discontinuing Study Drug Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants that had study drug discontinued regardless of study completion status was summarized.
Time Frame: Up to 4 weeks
Population: All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo
Number analyzed (Participants) | 16 | 5
Percentage of Participants | 0.0 | 40.0

11. Secondary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve of MK-2060 From 0 to Infinity (AUC0-inf)
Description: Plasma samples were collected at pre-specified time points post-dose and AUC0-inf was assessed.
Time Frame: Predose Day 1 and 1, 12, 24, 48, 52, 96, 168 hours postdose, then Days 12, 15, 22, 29, 60, 90, 120, 150
Population: Per-Protocol Population which consisted of the set of data generated by the subset of participants who had evaluable data for the endpoint and who complied with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/Liter
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg)
Number analyzed (Participants) | 6 | 7 | 6
hr*nmol/Liter | 4550 (61.2) | 6520 (63.4) | 15100 (31.7)
Statistical Analysis 1: Comparison: Part 1: Panel A- MK-2060 (8 mg); Test type: Other — Geometric mean ratio (GMR) was derived using the geometric mean (GM) for participants with ESRD and the GM from historical data obtained from a study of MK-2060 in healthy participants (PN001); GMR = 0.80, 90% CI 2-sided [0.54 to 1.18] — GMR=GM ESRD/GM Healthy
Statistical Analysis 2: Comparison: Part 1: Panel B- MK-2060 (20 mg); Test type: Other — GMR was derived using GM for participants with ESRD and the GM from historical data obtained from a study of MK-2060 in healthy participants (PN001); GMR = 0.53, 90% CI 2-sided [0.37 to 0.76] — GMR=GM ESRD/GM Healthy
Statistical Analysis 3: Comparison: Part 1: Panel A- MK-2060 (40 mg); GMR was derived using GM for participants with ESRD and the GM from historical data obtained from a study of MK-2060 in healthy participants (PN001); Test type: Other; GMR = 0.82, 90% CI 2-sided [0.55 to 1.21] — GMR=GM ESRD/GM Healthy

12. Secondary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve of MK-2060 From Time 0 to 168 Hours (AUC0-168)
Description: Plasma samples were collected at pre-specified time points post-dose and AUC0-168 hours was assessed.
Time Frame: Predose Day 1 and 1, 12, 24, 48, 52, 96, 168 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/Liter
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg)
Number analyzed (Participants) | 5 | 7 | 6
hr*nmol/Liter | 1560 (32.5) | 2420 (47.0) | 4930 (26.8)
Statistical Analysis 1: Comparison: Part 1: Panel A- MK-2060 (8 mg); [analysis description as in outcome 11, analysis 3]; Test type: Other; GMR = 1.41, 90% CI 2-sided [1.07 to 1.85] — GMR=GM ESRD/GM Healthy
Statistical Analysis 2: Comparison: Part 1: Panel B- MK-2060 (20 mg); [analysis description as in outcome 11, analysis 3]; Test type: Other; GMR = 0.86, 90% CI 2-sided [0.67 to 1.11] — GMR=GM ESRD/GM Healthy
Statistical Analysis 3: Comparison: Part 1: Panel A- MK-2060 (40 mg); [analysis description as in outcome 11, analysis 3]; Test type: Other; GMR = 0.82, 90% CI 2-sided [0.62 to 1.08] — GMR=GM ESRD/GM Healthy

13. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of MK-2060
Description: Plasma samples were collected at pre-specified time points post-dose and Cmax was assessed.
Time Frame: Predose Day 1 and 1, 12, 24, 48, 52, 96, 168 hours postdose, then Days 12, 15, 22, 29, 60, 90, 120, 150
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/Liter
Groups:
- Part 1: Panel A- MK-2060 (20 mg): Participants received a single 20-mg dose of MK-2060 via IV infusion
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel A- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg)
Number analyzed (Participants) | 6 | 7 | 6
nmol/Liter | 14.8 (38.2) | 28.0 (49.3) | 61.3 (19.3)
Statistical Analysis 1: Comparison: Part 1: Panel A- MK-2060 (8 mg); [analysis description as in outcome 11, analysis 3]; Test type: Other; GMR = 1.11, 90% CI 2-sided [0.84 to 1.46] — GMR=GM ESRD/GM Healthy
Statistical Analysis 2: Comparison: Part 1: Panel A- MK-2060 (20 mg); [analysis description as in outcome 11, analysis 3]; Test type: Other; GMR = 0.68, 90% CI 2-sided [0.52 to 0.87] — GMR=GM ESRD/GM Healthy
Statistical Analysis 3: Comparison: Part 1: Panel A- MK-2060 (40 mg); [analysis description as in outcome 11, analysis 3]; Test type: Other; GMR = 0.78, 90% CI 2-sided [0.60 to 1.03] — GMR=GM ESRD/GM Healthy

14. Secondary Outcome: Part 1: Plasma Concentration of MK-2060 at 168 Hours (C168)
Description: Plasma samples were collected at 168 hours post-dose and C168 was assessed.
Time Frame: 168 hours post dose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/Liter
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel A- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg)
Number analyzed (Participants) | 5 | 7 | 6
nmol/Liter | 6.29 (41.6) | 9.10 (57.7) | 15.8 (30.2)
Statistical Analysis 1: Comparison: Part 1: Panel A- MK-2060 (8 mg); [analysis description as in outcome 11, analysis 3]; Test type: Other; GMR = 1.50, 90% CI 2-sided [1.05 to 2.14] — GMR=GM ESRD/GM Healthy
Statistical Analysis 2: Comparison: Part 1: Panel A- MK-2060 (20 mg); [analysis description as in outcome 11, analysis 3]; Test type: Other; GMR = 0.91, 90% CI 2-sided [0.67 to 1.25] — GMR=GM ESRD/GM Healthy
Statistical Analysis 3: Comparison: Part 1: Panel A- MK-2060 (40 mg); [analysis description as in outcome 11, analysis 3]; Test type: Other; GMR = 0.86, 90% CI 2-sided [0.62 to 1.20] — GMR=GM ESRD/GM Healthy

15. Secondary Outcome: Part 1: Time to Maximum Observed Plasma Drug Concentration (Tmax) of MK-2060
Description: Plasma samples were collected at pre-specified time points post-dose and Tmax was assessed.
Time Frame: Predose Day 1 and 1, 12, 24, 48, 52, 96, 168 hours postdose
Population: as for outcome 11
Measure: Median (Full Range); unit: Hours
Groups:
- Part 1: Panel A- MK-2060 (40 mg): Participants received a single 8-mg dose of MK-2060 via IV infusion
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel A- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg)
Number analyzed (Participants) | 6 | 7 | 6
Hours | 1.13 [0.75 to 12.00] | 0.97 [0.83 to 12.00] | 1.09 [0.90 to 12.00]

16. Secondary Outcome: Part 1: Plasma Elimination Terminal Half-life (t ½) of MK-2060
Description: Plasma samples was collected at pre-specified time points post-dose and t ½ was assessed.
Time Frame: Predose Day 1 and 1, 12, 24, 48, 52, 96, 168 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel A- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg)
Number analyzed (Participants) | 6 | 7 | 6
Hours | 325 (88.5) | 422 (69.0) | 508 (21.7)

17. Secondary Outcome: Part 1: Plasma Clearance (CL) of MK-2060
Description: Plasma samples were collected at pre-specified time points post-dose and CL was assessed.
Time Frame: Predose Day 1 and 1, 12, 24, 48, 52, 96, 168 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel A- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg)
Number analyzed (Participants) | 6 | 7 | 6
Liters/hour | 0.0119 (61.2) | 0.0207 (63.4) | 0.0179 (31.7)

18. Secondary Outcome: Part 1: Plasma Volume of Distribution (Vz) of MK-2060
Description: Plasma samples were collected at pre-specified time points post-dose and Vz was assessed.
Time Frame: Predose Day 1 and 1, 12, 24, 48, 52, 96, 168 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel A- MK-2060 (20 mg) | Part 1: Panel A- MK-2060 (40 mg)
Number analyzed (Participants) | 6 | 7 | 6
Liters | 5.56 (49.0) | 12.6 (65.3) | 13.1 (31.2)

19. Secondary Outcome: Part 2: AUC0-168 of MK-2060
Description: Plasma samples were collected at pre-specified time points post-dose and AUC0-168 hours was assessed.
Time Frame: Up to 168 hours on Day 1 and Day 22
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/L
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance
Number analyzed (Participants) | 15
hr*nmol/L
  Day 1: number analyzed (Participants) | 11
  Day 1 | 2290 (26.8)
  Day 22 | 9880 (28.9)

20. Secondary Outcome: Part 2: Cmax of MK-2060
Description: Plasma samples were collected at pre-specified time points post-dose and Cmax was assessed.
Time Frame: Day 1 and Day 22
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/Liter
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance
Number analyzed (Participants) | 16
nmol/Liter
  Day 1: number analyzed (Participants) | 15
  Day 1 | 32.6 (32.5)
  Day 22 | 90.9 (30.4)

21. Secondary Outcome: Part 2: C168 of MK-2060
Description: Plasma samples were collected at 168 hours post-dose and C168 was assessed.
Time Frame: 168 hours post dose on Days 1 and 22
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/Liter
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance
Number analyzed (Participants) | 15
nmol/Liter
  Day 1: number analyzed (Participants) | 11
  Day 1 | 54.1 (42.1)
  Day 22 | 43.8 (30.5)

22. Secondary Outcome: Part 2: Tmax of MK-2060
Description: Plasma samples were collected at pre-specified time points post-dose and Tmax was assessed.
Time Frame: Day 1 and Day 22
Population: as for outcome 11
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance
Number analyzed (Participants) | 16
Hours
  Day 1 | 1.00 [0.92 to 47.92]
  Day 22: number analyzed (Participants) | 15
  Day 22 | 1.00 [0.00 to 24.00]

23. Secondary Outcome: Fold Change From Baseline in Activated Partial Thromboplastin Time (aPTT) of MK-2060: Part 1
Description: Plasma samples were collected at pre-specified time points post-dose and aPTT values were assessed. The fold change (Day 8/Baseline) at Day 8 was reported.
Time Frame: Baseline and 168 hours post-dose (Day 8)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel A- MK-2060 (20 mg) | Part 1: Panel C- MK-2060 (40 mg) | Part 1: Placebo
Number analyzed (Participants) | 5 | 7 | 6 | 5
Ratio | 1.04 [0.92 to 1.18] | 1.17 [1.06 to 1.30] | 1.52 [1.36 to 1.71] | 1.05 [0.92 to 1.19]

24. Secondary Outcome: Fold Change From Baseline in aPTT of MK-2060: Part 2
Description: as for outcome 23
Time Frame: Baseline and Day 8
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo
Number analyzed (Participants) | 15 | 4
Ratio | 2.46 [1.95 to 3.11] | 0.68 [0.43 to 1.06]

ADVERSE EVENTS:
Time Frame: Up to 164 days
Description: Analysis population was the All Subjects as Treated Population which consisted of all participants who received at least one dose of treatment.
Arm/Group | Part 1: Panel A- MK-2060 (8 mg) | Part 1: Panel B- MK-2060 (20 mg) | Part 1: Panel C- MK-2060 (40 mg) | Part 1: Placebo | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/5 | 0/16 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 1/6 | 0/5 | 1/16 | 3/5
Other Adverse Events (participants affected / at risk) | 1/6 | 4/7 | 3/6 | 3/5 | 1/16 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Panel A- MK-2060 (8 mg) (N=6) | Part 1: Panel B- MK-2060 (20 mg) (N=7) | Part 1: Panel C- MK-2060 (40 mg) (N=6) | Part 1: Placebo (N=5) | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance (N=16) | Part 2: Placebo (N=5)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Panel A- MK-2060 (8 mg) (N=6) | Part 1: Panel B- MK-2060 (20 mg) (N=7) | Part 1: Panel C- MK-2060 (40 mg) (N=6) | Part 1: Placebo (N=5) | Part 2: MK-2060 25-mg Loading/ 25-mg Maintenance (N=16) | Part 2: Placebo (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. The Sponsor will comply with the requirements for publication of study results. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT03873038/Prot_SAP_000.pdf